CLINICAL TRIAL: NCT06434012
Title: Barts Endocarditis Research Registry
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 249740
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Infective Endocarditis; Endocarditis; Endocarditis, Bacterial
MeSH Terms: conditions — Endocarditis; Endocarditis, Bacterial | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: registry — This is registry for Infective Endocarditis

SUMMARY:
The Barts Endocarditis Research Registry is being set up to give a unique opportunity to assess the characteristics of Infective Endocarditis (IE) in our population cohort, the current use of imaging techniques, as well as the implementation of the ESC guidelines and its consequence in terms of prognosis. All this will help improve the diagnosis and management of IE. The registry will also form the core of all our subsequent work, including interventional studies. The endocarditis research registry is to record the epidemiological, demographic, microbiological, surgical and outcome data in our cohort of endocarditis patients. This work will underpin all future work in endocarditis by clearly defining our patient cohort and the outcomes from treatment. We have a series of studies planned that we believe will influence the management of endocarditis (we are working up proposals for genomic and therapeutic trials that will subsequently be presented for ethical and hospital approval). The registry will be generic to all our planned studies, and will allow us to capture data to assess treatment effectiveness

DETAILED DESCRIPTION:
This research registry will give us the unique opportunity to assess the characteristics of IE in our population cohort, the current use of imaging techniques, as well as the implementation of the ESC guidelines and its consequence in terms of prognosis. All this will help improve the diagnosis and management of IE. The registry will also form the core of all our subsequent work, including interventional studies.

Infective endocarditis (IE) is a rare but serious disease, associated with high morbidity and in-hospital mortality. Despite improvements in diagnostic and therapeutic strategies the mortality remains at 15-30% in most published studies. The reasons for this persistent poor prognosis are numerous and include older patients with more severe disease, changes in the epidemiologic profiles and more patients with prosthetic or device related IE.

Following the formation of Barts Heart Centre (BHC) there was a sharp and noticeable increase in the number of patients with infective endocarditis (IE) referred to our centre. Recognising this change, the complexity of patients, and the coincident publication of the European Society of Cardiology Guidelines on Infective Endocarditis (2015), our Specialised Cardiology Directorate set up a new referral pathway, Standard Operating Procedure and Endocarditis Team meeting (MDT). The aim was to ensure focussed, consistent, and evidence-based care with joint medical and surgical input to this unique group of very unwell patients, with high inpatient mortality. In addition, the MDT would discuss and co-ordinate the care of all IE patients, with a weekly discussion of those on site, as well as at our referring hospitals. The MDT started in October 2015 and is composed of representatives from Cardiology (including imaging), Cardiac Surgery, Microbiology, Radiology/Nuclear Medicine and Pharmacy.

Since its inception, the MDT has discussed 367 patients at BHC and our wider referral centres (October 2015 - January 2018). Of those patients, 298 have been confirmed/probable as having IE: 144 surgically managed; 139 medically managed; 16 device extractions with intracardiac infection, all following international guidance. This does not include the grown-up congenital heart disease patients who are discussed and managed separately.

An audit database to track outcomes was started in January 2018, but there is a need to expand this work and make a registry that will form the foundation of all other research that we will undertake.

Mortality across the cohort has been at the lower end of international publications at 17.1% (51/298). Our current surgical mortality stands at 4.7% (14/298), which represents a significant reduction compared to pre-merger where combined mortality at the individual hospitals was 12.2%. In those patients who have died with medical management (37/51), the vast majority have had advanced life-limiting non-cardiac co-morbidities that preclude cardiac surgery (n=19) or on-going intravenous drug use after previous cardiac surgery for IE (n=6). Six patients have not been referred in time for surgery, having presented locally with septic shock and deteriorated rapidly, and this is an area of further education for our referring centres. Six patients have had operations without intra-operative evidence of infection. However, these patients had indications for surgery due to haemodynamically significant regurgitant valve disease.

Our morbidity and mortality reviews have allowed us to learn from all these cases, across all specialties and imaging modalities.

Not only has this approach led to improvements in patient care, but it has also raised the profile of BHC as a centre of special expertise. Our referring centres now include the DGH's of Barts Health NHS Trust (Whipps Cross University Hospital, Newham University Hospital, and The Royal London Hospital), plus many other district general hospitals in our locale.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged 16 and over (Patients under 16 years of age are not admitted to Barts Heart Centre)

  * Patients admitted to Barts Heart Centre with confirmed Endocarditis (see above)
  * Patients attending outpatients with confirmed/suspected Endocarditis
  * Patients with possible IE who complete treatment for endocarditis
  * Patients with cardiac device related Endocarditis
  * Patients with the ability to provide informed consent

Exclusion Criteria:

* • Patients with pacemaker pocket infection with no evidence of pacemaker lead or valve infection

  * Patients who refuse consent to be included in the research database
  * Patients with "rejected" endocarditis

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: There are approximately 150 cases of endocarditis each year treated within the trust and recruitment is expected to be rapid
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2029-04-24 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
To define current mortality rates for patients treated for endocarditis at Barts Heart Centre | 10 years
  The primary goal of the endocarditis registry is to record the epidemiological, demographic, microbiological, surgical and outcome data in our cohort of endocarditis patients. This work will underpin all future work in endocarditis by clearly defining our patient cohort and the outcomes from treatment.
To define current morbidity rates for patients treated for endocarditis at Barts Heart Centre | 10 years
  The primary goal of the endocarditis registry is to record the epidemiological, demographic, microbiological, surgical and outcome data in our cohort of endocarditis patients. This work will underpin all future work in endocarditis by clearly defining our patient cohort and the outcomes from treatment.
To define current rates of reinfection for patients treated for endocarditis at Barts Heart Centre | 10 years
  The primary goal of the endocarditis registry is to record the epidemiological, demographic, microbiological, surgical and outcome data in our cohort of endocarditis patients. This work will underpin all future work in endocarditis by clearly defining our patient cohort and the outcomes from treatment.
To define current rates of relapse for patients treated for endocarditis at Barts Heart Centre | 10 years
  The primary goal of the endocarditis registry is to record the epidemiological, demographic, microbiological, surgical and outcome data in our cohort of endocarditis patients. This work will underpin all future work in endocarditis by clearly defining our patient cohort and the outcomes from treatment.

SECONDARY OUTCOMES:
To collect data regarding infecting organism, valve appearances and pathological markers and investigate their relationship to mortality, morbidity, reinfection and relapse rates | 10 years
  A secondary aim will be to use the registry to develop a series of observational studies, especially how the infecting organism interacts with the diagnostic indices in our labs and imaging protocols
To collect data regarding infecting organism and investigate its relationship to mortality, morbidity, reinfection and relapse rates | 10 years
  A secondary aim will be to use the registry to develop a series of observational studies, especially how the infecting organism interacts with the diagnostic indices in our labs and imaging protocols
To collect data regarding valve appearance and investigate its relationship to mortality, morbidity, reinfection and relapse rates | 10 years
  A secondary aim will be to use the registry to develop a series of observational studies, especially how the infecting organism interacts with the diagnostic indices in our labs and imaging protocols
To collect data regarding pathological markers and investigate its relationship to mortality, morbidity, reinfection and relapse rates | 10 years
  A secondary aim will be to use the registry to develop a series of observational studies, especially how the infecting organism interacts with the diagnostic indices in our labs and imaging protocols

CONTACTS AND LOCATIONS:
Overall Officials: Simon Woldman, MSc, Principal Investigator — St Bartholomews Hospital
Locations (1):
- St Bartholomews Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided